CLINICAL TRIAL: NCT04785807
Title: STRESS From in Charge Relative Facing the Announcement of Decisions Limiting or Stopping Treatments in Emergency Room During the COVID-19 Epidemic
Acronym: COVER ACC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 69HCL20_0678
Record Dates: First submitted 2021-02-23; First posted 2021-03-08 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Covid19; Post Traumatic Stress Disorder; Anxiety
Keywords: HADS; IES-R; Family; Limitation or discontinuation of treatment
MeSH Terms: conditions — COVID-19; Stress Disorders, Post-Traumatic; Anxiety Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluation arm (Experimental)
  Interventions: Other: Post traumatic, Anxiety and depression evaluation

INTERVENTIONS:
Other: Post traumatic, Anxiety and depression evaluation — Family member of person or trust of patient who had a limitation or discontinuation of treatments will be identified and asked to fulfilled a hospitalized anxiety and depression scale and the revised Impact Event scale 7 and 30 days after the limitation or discontinuation of treatments announcement

SUMMARY:
In the context of the COVID-19 pandemic, the emergency reception services had to be radically reorganized. In this tense environment, professionals must face ethical dilemmas, make referral decisions and prioritize patients. Due to the limited number of visits to many hospitals, interactions with relatives and families of patients are mainly conducted by phone. These limitations will continue as long as the context of uncertainty over the course of the pandemic persists. Limitation or discontinuation of treatment (LDT) announcements were therefore also impacted and the exceptional situation related to COVID-19 reinforces the difficulties encountered by professionals in usual time (place of announcement, inappropriate lack of time, etc.). Thus, LDTs are most often done over the phone without the families being able to go to the hospital. Because of this, these announcements can be more traumatic. Investigators have already highlighted in a recent study the lack of communication between caregivers and families in the context of LDT announcements and the context of COVID 19 exacerbated these aspects given the limitations of visits.

The investigators therefore propose to study the experiences of families who are notified of a decision to limit or stop treatment by phone in the emergency room during the COVID-19 crisis.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old.
* Person of trust designated in writing or contact person if designated by the family or primary caregiver or failing that the family member or person of trust of an adult patient deemed unfit to receive the information (advanced dementia (lower MMS) to 10), disturbance of consciousness). Only one person per family will be included.
* having been informed of a LAT decision in the emergency room by telephone during the pandemic
* Having consented to participate in the study
* Affiliated with social security

Exclusion Criteria:

* Person of trust, family or close friend unable to understand or write in French.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-03-30 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Post traumatic syndrome evaluated thanks to the Revised impact event scale (IES-R) | 30 days after limitation or discontinuation of treatment announcement
  The primary endpoint is the evaluation of Post traumatic syndrome among the family member or person of trust of a patient who received a limitation or discontinuation of treatment, 30 days after this announcement. The post traumatic syndrome will be evaluated thanks to the Revised impact event scale (IES-R) giving a score going from 0 to 88. The greater the score, the worse the outcome is.

SECONDARY OUTCOMES:
Anxiety level at day 7, assessed using the Hospitalized Anxiety and Depression Scale-(HADS) | 7 days after inclusion
  Evaluation of Anxiety among the family member or person of trust of a patient who received a limitation or discontinuation of treatment, 7 days after this announcement. Anxiety will be assessed using the Hospitalized Anxiety and Depression Scale, giving two scores (one for anxiety, one for depression) going from 0 to 21. The greater the score, the worse the outcome is.
Depression level at day 7, assessed using the Hospitalized Anxiety and Depression Scale | 7 days after inclusion
  Evaluation of Depression among the family member or person of trust of a patient who received a limitation or discontinuation of treatment 7 days after this announcement, using the Hospitalized Anxiety and Depression Scale, giving two scores (one for anxiety, one for depression) going from 0 to 21. The greater the score, the worse the outcome is.
Anxiety level at day 30, assessed using the Hospitalized Anxiety and Depression Scale (HADS) | 30 days after inclusion
  Evaluation of Anxiety among the family member or person of trust of a patient who received a limitation or discontinuation of treatment 30 days after this announcement, using the Hospitalized Anxiety and Depression Scale, giving two scores (one for anxiety, one for depression) going from 0 to 21. The greater the score, the worse the outcome is.
Depression level at day 30, assessed using the Hospitalized Anxiety and Depression Scale (HADS) | 30 days after inclusion
  Evaluation of Depression among the family member or person of trust of a patient who received a limitation or discontinuation of treatment, 30 days after this announcement. Anxiety will be assessed using the Hospitalized Anxiety and Depression Scale, giving two scores (one for anxiety, one for depression) going from 0 to 21. The greater the score, the worse the outcome is.
Description of socio-demographic factors | 30 days after inclusion
  In order to determine anxiety and depression risk factors, the individual socio-demographic factors such as recourse to psychological support, consumption of psychoactive substances (caffeine, tobacco, psychotropic drugs, anxiolytics) will be described.
Description of clinical factors | 30 days after inclusion
  In order to determine anxiety and depression risk factors, the factors linked to the patient (COVID infection, death) will be described.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Service des urgences, Hôpital Edouard Herriot, Hospices Civils de Lyon, Lyon
  - service des urgences, Hôpital de la Croix-Rousse, Hospices Civils de Lyon, Lyon
  - Service d'Accueil des Urgences, Hôpital Lyon Sud, Hospices Civils de Lyon, Pierre-Bénite